CLINICAL TRIAL: NCT01324492
Title: A Phase Ib, Open-label Study to Evaluate RAD001 as Monotherapy Treatment in Chinese Patients With Advanced Pulmonary Neuroendocrine Tumor
Brief Title: Safety and Efficacy of RAD001 in Chinese Patients With Advanced Pulmonary Neuroendocrine Tumor
Acronym: \MACS1304
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001KCN01
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Lung Neuroendocrine Neoplasm
Keywords: phase Ib,; RAD001,; advanced pulmonary neuroendocrine tumor
MeSH Terms: interventions — Everolimus

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001
  Other Names: Everolimus

SUMMARY:
The present study is designed to collect safety/tolerability data and explore the efficacy of RAD001 in advanced pulmonary neuroendocrine tumor in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoid tumors
* Newly diagnosed advanced carcinoid tumors or progressed after 1st line treatment is eligible

Exclusion Criteria:

* Patients with either clinically apparent central nervous system metastases or carcinomatous meningitis(non-clinical symptoms with brain lesions is eligible)
* Received Cytotoxic chemotherapy, immunotherapy or radiotherapy prior to enrollment
* Patients with a concurrent malignancy, or history of prior malignancy within the past three years, except for basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, treated early stage (T1a) prostate cancer or treated early stage (DCIS or LCIS) breast cancer
* Prior therapy with RAD001 or other mTOR inhibitors (sirolimus, temsirolimus, everolimus)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adverse events, serious adverse events, laboratory results (Hematology, Serum Blood Chemistry, hepatitis tests, Standard urinalysis dipstick assessment, Coagulation Studies)or assessment of the incidence of pneumonitis | every 6 weeks

SECONDARY OUTCOMES:
Chest X-Ray,Triphasic CT scan or MRI of the chest, abdomen and cavitas pelvis evaluated by using RECIST criteria | 6 weeks
Date and reason of death, or discontinuation from the study. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Investigative Site
Locations (4):
- China (4):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning